CLINICAL TRIAL: NCT06690853
Title: Effects of Coordinative Warm-Up Exercise Protocols on the Technical and Cognitive Performance of Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Collaborators: Marco Centorbi (Unknown); Alessandra di Cagno (Unknown); Giuseppe Calcagno (Unknown); Andrea Buonsenso (Unknown)
Responsible Party: Principal Investigator, Giovanni Fiorilli, Principal Investigator, University of Molise
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25/2023
Record Dates: First submitted 2024-11-09; First posted 2024-11-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Soccer Performance
Keywords: soccer players; warm up; technical-coordination; cortisol; adrenaline; noradrenaline; dopamine; football
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental coordinative training (Experimental): The warm-up protocols of the Experimental Group included four types of upper and lower limb coordination exercises using different-sized balls, with intensity increasing week by week. The warm-up exercises were conducted four times per week, including game day, for a total of 12 weeks.
  Interventions: Other: Experimental Coordinative training
- Traditional training (control group) (Active Comparator): The Control Group warm-up protocol only involved joint mobility exercises and muscle activation, as used in their regular training activities.
  Interventions: Other: Traditional training (control group)

INTERVENTIONS:
Other: Experimental Coordinative training — The warm-up protocols of the Experimental Group included four types of upper and lower limb coordination exercises using different-sized balls, with intensity increasing week by week.
  Arms: experimental coordinative training
Other: Traditional training (control group) — The Control Group warm-up protocol only involved joint mobility exercises and muscle activation, as used in their regular training activities.
  Arms: Traditional training (control group)

SUMMARY:
The aim of this study is to evaluate the effects of 12 weeks of warm-up protocols administered to elite soccer players on technical-coordination performance and levels of cortisol, adrenaline, noradrenaline, and dopamine, measured before and after the intervention.

DETAILED DESCRIPTION:
The warm-up protocols included coordination exercises using different types of balls, with combined activities involving both the upper and lower limbs

ELIGIBILITY:
Inclusion Criteria:

* elite soccer players

Exclusion Criteria:

* no injuries in the previous 6 months;
* no adherence to other training protocols;
* no use of prohibited drugs and/or supplements that could affect the test results and exercises

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Illinois agility test | at 12 weeks
  Illinois Test with the ball, aiming to achieve the best time to complete the test.
Illinois agility test | at 12 weeks
  Illinois Test without the Ball, aiming to achieve the best time to complete the test
agility test | at 12 weeks
  Planned Y Test (right and left), aiming to achieve the best time to complete the test
agility test | at 12 weeks
  Unplanned Y Test (right and left), aiming to achieve the best time to complete the test
Loughborough Soccer Shooting Test | at 12 weeks
  Right and Left Side Shooting Accuracy Test.
Blood analysis | at 12 weeks
  adrenaline
Blood analysis | at 12 weeks
  noradrenaline
Blood analysis | at 12 weeks
  cortisol
Blood analysis | at 12 weeks
  dopamine

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi del Molise, Campobasso, CB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Centorbi M, Medoro A, Modolo L, Di Claudio G, Di Martino G, Della Valle C, Buonsenso A, Marziliano N, Davinelli S, Calcagno G, di Cagno A, Fiorilli G. Reactive Training in Enhancing Technical Performance and Modulating Cortisol Biomarkers in Competitive Soccer Players. J Strength Cond Res. 2026 Jan 28. doi: 10.1519/JSC.0000000000005390. Online ahead of print. PMID 41591377